CLINICAL TRIAL: NCT02753907
Title: Impact of an 8-week Linoleic Acid Intake in Soy Oil on Lp-PLA2 Activity in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LA_fu
Record Dates: First submitted 2016-04-22; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Healthy Subjects

ARMS (3):
- Low LA (linoleic acid) (Experimental): Individuals who replaced 10 mL soy oil with one apple
  Interventions: Dietary Supplement: Low LA
- Medium LA (No Intervention): Individuals who maintained their usual food intake
- High LA (Experimental): Individuals who reduced 1/3 cup of cooked refined rice and consumed 9.9 g of soy oil as a supplement
  Interventions: Dietary Supplement: High LA

INTERVENTIONS:
Dietary Supplement: Low LA — Individuals who replaced 10 mL soy oil with one apple
  Arms: Low LA (linoleic acid)
Dietary Supplement: High LA — Individuals who reduced 1/3 cup of cooked refined rice and consumed 9.9g (9 of 1.1g capsules, 3 capsules at every 3 meals a day) of soy oil as a supplement
  Arms: High LA

SUMMARY:
Self-reported healthy participants (n=150) aged 30-65 years with 18.5 kg/m^2 ≤ BMI < 30 kg/m^2 were randomly assigned into three groups: a low linoleic acid (LA, 18:2n-6) group (n=50) replaced 10 mL soy oil with one apple; a medium LA group (control group, n=50) maintained usual food intake; a high LA group (n=50) reduced 1/3 cup of cooked refined rice and consumed 9.9g of soy oil capsules daily as a supplement. Plasma fatty acids and lipoprotein-associated phospholipase A2 (Lp-PLA2) activity were measured at baseline and 8 week alongside other cardiovascular disease risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 65 years at beginning of study
* Subjects with BMI 18.5 to 30 kg/m^2

Exclusion Criteria:

* Use of any medication or supplements that alter lipid metabolism.
* Presence of dyslipidemia, diabetes mellitus, hypertension, liver disease, renal disease, chronic disease of the gastrointestinal tract, cerebrovascular disease, pancreatitis or cancer.
* Women who pregnant or lactating.
* Drug or alcohol abuse.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in Lp-PLA2 activity (nmol/mL/min) | At baseline and end of each 8-week diet period

SECONDARY OUTCOMES:
Change in total cholesterol (mg/dL) | At baseline and end of each 8-week diet period
Change in LDL cholesterol (mg/dL) | At baseline and end of each 8-week diet period
  Lipids and lipoproteins, such as total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, Apo A-I, Apo B
Change in HDL cholesterol (mg/dL) | At baseline and end of each 8-week diet period
Change in triglyceride (mg/dL) | At baseline and end of each 8-week diet period

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomics, Yonsei University., Seoul, South Korea

REFERENCES:
- [Derived] Kim M, Kim M, Lee A, Yoo HJ, Her JS, Jee SH, Lee JH. Impact of 8-week linoleic acid intake in soy oil on Lp-PLA2 activity in healthy adults. Nutr Metab (Lond). 2017 May 8;14:32. doi: 10.1186/s12986-017-0186-2. eCollection 2017. PMID 28503188